CLINICAL TRIAL: NCT03369977
Title: Multi-center, Randomized, Controlled Clinical Trial of BioGlue Surgical Adhesive as an Adjunct for Structural Repair and Hemostasis in Chinese Patients With Acute Type A Aortic Dissections.
Brief Title: BioGlue as an Adjunct for Structural Repair and Hemostasis in Chinese Acute Type A Aortic Dissections Patients
Acronym: CHINA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CryoLife, Inc. (Industry)
Responsible Party: Sponsor
Organization: CryoLife (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIO1601.000-C(10/16)
Record Dates: First submitted 2017-11-30; First posted 2017-12-12 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Type A Aortic Dissection
Keywords: BioGlue Surgical Adhesive; Type A Aortic Dissection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- BioGlue Surgical Adhesive (Experimental): Subjects in the BioGlue group will receive BioGlue as an adjunct for traditional surgical repair of the sinus of Valsalva.
  Interventions: Device: BioGlue Surgical Adhesive
- Traditional Surgical Repair (Other): Subjects in the control group will receive traditional surgical repair of the sinus of Valsalva.
  Interventions: Other: Traditional Surgical Repair

INTERVENTIONS:
Device: BioGlue Surgical Adhesive — BioGlue (produced by CryoLife in Kennesaw, GA) is a surgical adhesive with two components respectively purified bovine serum albumin (BSA) and Glutaraldehyde (their proportions are 4:1). Crosslinked bonds (covalent bonds) of Glutaraldehyde cross-link the protein on the surface of the tissue and the amino residue of the bovine serum albumin. BioGlue also adheres to the synthetic matrix material by a mechanical interlocking mechanism in the space of graft matrix.
  Arms: BioGlue Surgical Adhesive
Other: Traditional Surgical Repair — Traditional surgical repair as determined by the surgeon
  Arms: Traditional Surgical Repair

SUMMARY:
A multi-center, randomized, controlled clinical trial is designed to investigate the safety and efficacy of BioGlue as an adjunct for structural repair and hemostasis to traditional surgical repair in Chinese subject with Acute type A aortic dissections.

DETAILED DESCRIPTION:
A multi-center, randomized, controlled clinical trial is designed to investigate the safety and efficacy of BioGlue as an adjunct for structural repair and hemostasis in Chinese subjects with acute type A aortic dissection. The trial consists of three phases:

Phase One - A non-randomized, lead-in phase. During the lead-in phase, the first 2-3 eligible subjects at each center will receive BioGlue in open surgery. These subjects will be evaluated for safety separately from the randomized phase of the trial.

Phase Two - A randomized, controlled phase. Type A aortic dissection subjects will be randomized into TSR group (control group) and surgical repair with BioGlue group (test group) with a ratio of 1:1, so that equal number of subjects in test and control groups can be ensured.

Phase Three - A Follow-up of Late Safety Outcomes of using BioGlue in "The CHINA Trial" . Subjects enrolled in "The CHINA Trial," from both the BioGlue and the control (TSR) group, will be invited to participate. Clinical data evaluating mortality, adverse events, and re-operation rates will be collected from subject's medical charts.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18-70 years of age.
* Subject has a confirmed diagnosis of acute type A aortic dissection with subtype A2.
* Subject is willing and able to give written consent for the trial. If the subject is unconscious or under the influence of medications which render him or her unable to give fully informed consent, a guardian may provide informed consent for the subject regarding trial participation.

Exclusion Criteria:

* Subjects with known allergy to albumin, bovine products, or glutaraldehyde.
* Subjects who have been treated with an investigational product who have not completed the entire follow-up period.
* Subjects who do not meet the eligibility criteria, including those who do not wish to participate or give informed consent for trial participation, will not be enrolled into the trial, and will be offered equivalent, non-trial surgical or other treatment, as judged appropriate by the investigator.
* Subjects with previous cardiac and aortic surgery.
* End stage malperfusion syndromes (i.e. end-organ failure such as coma, paraplegia, hemiplegia, intestinal necrosis, or hepatic failure).
* Subjects with Marfan syndrome or other connective tissue disorders.
* Previous chronic dissections resulting from non-cardiac surgery and/or trauma.
* Concomitant surgery of valve replacement (both in screening and intraoperative).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-06-24 (Actual); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Successful Closure of the False Lumen | This success can be visually confirmed intraoperatively with a TEE (binary yes/no expression for each subject)
  Successful closure of the false lumen as determined by intraoperative TEE. With successful closure of the false lumen, a complete disappearance of the false lumen will be achieved.

SECONDARY OUTCOMES:
Successful closure of the false lumen by CTA or TTE at discharge | CTA or TTE scan at discharge or at 20 days (+/- 10 days) post-operatively for subjects with longer hospital stays.
  Successful closure of the false lumen at discharge or at 20 days (+/- 10 days) post-operatively confirmed by CTA scan or Transthoracic Echocardiogram (TTE) scan if the subject is unable to have a CTA.
Time to repair the sinuses of Valsalva | The time for repairing the sinuses of Valsalva will be documented intraoperatively.
  During the operation the time to repair the sinuses of Valsalva will be recorded.
Evaluate the successful hemostasis at the anastomotic site | The measurement begins intraoperatively after either BioGlue or Traditional Surgical Repair is applied to the anastomotic suture line(s) and the bypass cross clamp is released.
  Hemostasis is assessed visually (i.e. lack of any observable extravascular bleeding) and is monitored until hemostasis is achieved at each applied anastomotic site.
Treatment failure of the aortic dissection repair site identified in "The CHINA Trial" which leads to either post-discharge mortality or re-operation. | The measurement begins at discharge and will end when the retrospective chart review is performed by the hospital (could be up to 3 years post-op)
  Post-operative mortality and re-operation(s) will be collected from the subjects' medical charts retrospectively and during informed consent telephone notification.
Proportion of subjects with device-related or procedure-related adverse events, determined by the investigators. | The measurement begins at discharge and will end when the retrospective chart review is performed by the hospital (could be up to 3 years post-op).
  Post-operative adverse event(s) will be collected from the subjects' medical charts retrospectively. Assessment will only be performed on the surgical site from "The CHINA Trial," defined as obliteration of the false lumen (BioGlue group) or repair of acute type A aortic dissection (control group) and anastomosis (both BioGlue and control groups).

CONTACTS AND LOCATIONS:
Overall Officials: Scott B Capps, MS, Study Director — CryoLife, Inc.
Locations (7):
- China (7):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing
  - Nanjing Drum Tower Hospital, The Affiliated Hospital of Nanjing University Medical School, Nanjing
  - Nanjing First Hospital, Nanjing
  - Changhai Hospital,The Second Military Medical University, Shanghai
  - Zhongshan Hospital, Fudan University, Shanghai
  - Wuhan Asia Heart Hospital, Wuhan
  - Henan Provincial People's Hospital, Zhengzhou